CLINICAL TRIAL: NCT01033409
Title: Comparative Phase I Safety and Immunogenicity in Adult Volunteers of Three Recombinant Attenuated Salmonella Typhi Vaccine Vectors Producing Streptococcus Pneumoniae Surface Protein Antigen PspA
Brief Title: Recombinant Attenuated Salmonella Typhi Vaccine Vectors Producing Streptococcus Pneumoniae PspA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 09-RASV-Sp-01
Record Dates: First submitted 2009-11-16; First posted 2009-12-16 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Pneumonia
Keywords: Salmonella Typhi; pneumonia; oral; vaccine
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S. Typhi-vectored pneumo vaccine 10^7 (Experimental): Arm 1 will evaluate three attenuated S. Typhi strains administered to 3 groups of 5 subjects in single oral doses (10^7 CFU) for safety and immunogenicity. Dose escalation for each strain will proceed after demonstrating the safety and tolerability of 10^7 CFU oral dosage through Day 28.
  Interventions: Biological: Salmonella Typhi-vectored pneumonia vaccine
- S. Typhi-vectored pneumo vaccine 10^8 (Experimental): Arm 2 will evaluate three attenuated S. Typhi strains administered to 3 groups of 5 subjects in single oral doses (10^8 CFU) for safety and immunogenicity. Dose escalation for each strain will proceed after demonstrating the safety and tolerability of 10^8 CFU oral dosage through Day 28.
  Interventions: Biological: Salmonella Typhi-vectored pneumonia vaccine
- S. Typhi-vectored pneumo vaccine 10^9 (Experimental): Arm 3 will evaluate three attenuated S. Typhi strains administered to 3 groups of 5 subjects in single oral doses (10^9 CFU) for safety and immunogenicity. Dose escalation for each strain will proceed after demonstrating the safety and tolerability of 10^9 CFU oral dosage through Day 28.
  Interventions: Biological: Salmonella Typhi-vectored pneumonia vaccine
- S. Typhi-vectored pneumo vaccine 10^10 (Experimental): Arm 4 will evaluate three attenuated S. Typhi strains administered to 3 groups of 5 subjects in single oral doses (10^10 CFU) for safety and immunogenicity. Dose escalation for each strain will proceed after demonstrating the safety and tolerability of 10^10 CFU oral dosage through Day 28.
  Interventions: Biological: Salmonella Typhi-vectored pneumonia vaccine

INTERVENTIONS:
Biological: Salmonella Typhi-vectored pneumonia vaccine — Liquid, oral dosage administered once at 10^7 CFU in 10 mL phosphate-buffered saline
  Other Names: RASV strains
  Arms: S. Typhi-vectored pneumo vaccine 10^7
Biological: Salmonella Typhi-vectored pneumonia vaccine — Liquid, oral dosage administered once at 10^8 CFU in 10 mL phosphate-buffered saline
  Other Names: RASV strains
  Arms: S. Typhi-vectored pneumo vaccine 10^8
Biological: Salmonella Typhi-vectored pneumonia vaccine — Liquid, oral dosage administered once at 10^9 CFU in 10 mL phosphate-buffered saline
  Other Names: RASV strains
  Arms: S. Typhi-vectored pneumo vaccine 10^9
Biological: Salmonella Typhi-vectored pneumonia vaccine — Liquid, oral dosage administered once at 10^10 CFU in 10 mL phosphate-buffered saline
  Other Names: RASV strains
  Arms: S. Typhi-vectored pneumo vaccine 10^10

SUMMARY:
In this Phase I clinical study, three recombinant, avirulent Salmonella Typhi (RASV) strains each expressing the Streptococcus pneumoniae surface protein, PspA, will be compared as live biological vaccine vectors to evaluate safe and tolerable, single, oral dose levels in adult subjects.

DETAILED DESCRIPTION:
The use of attenuated Salmonella strains that are unable to cause clinical disease but trigger a self-limiting infection leading to stimulation of protective immunity presents an attractive alternative to killed and subunit vaccines. Live, attenuated Salmonella strains have been shown to be excellent carriers, or vectors, for prokaryotic or eukaryotic antigens, being able to stimulate strong systemic and local immune responses against the expressed antigens. Three Salmonella Typhi strains have been engineered to express a gene encoding the alpha-helical domain of the Streptococcus pneumoniae surface protein, PspA, and will serve as live biological vaccine vectors in the proposed clinical trial to evaluate maximum safe and tolerable single dose levels after their oral administration to subjects. In this Phase I study, healthy young adults 18-40 years of age will participate in a dose escalating, dose sequential study divided into four Arms to receive doses of 10^7, 10^8, 10^9 and 10^10 CFU. Each Arm (1-4) will consist of 3 groups of 5 subjects per group to receive a single oral dose of one of three recombinant attenuated S. Typhi vaccine vectors producing the pneumococcal antigen PspA. Each group per Arm will receive the same dose of one of the three vaccines for a total of 60 subjects (15 subjects per dose-escalating Arm, 3 groups per Arm, 5 subjects per group). Subject participation lasts 6 months after receiving the oral vaccine dosage with approximately the first 12-15 days (study Days 0-14) in confinement. Release criteria include 2 negative blood cultures in a row through study Day 7 (inpatient monitoring for 8 days) and 2 negative stool cultures in a row through study Day 5. The objectives of the study are 1) to evaluate maximum safe tolerable single dose levels of the three recombinant attenuated S. Typhi vaccine vectors using dose-escalation, dose-sequential studies in healthy adult subjects, and 2) to evaluate immunogenicity of the three recombinant attenuated S. Typhi vaccine vectors with regard to their abilities to induce mucosal and systemic antibody responses to the S. pneumoniae PspA and S. Typhi antigens. The vaccines are not anticipated to prevent disease. Although the immune responses generated by the vaccine vectors may confer some degree of protection against future infection with S. pneumoniae and S. Typhi, such protection is incidental. It is not the goal of this study to develop or test either a pneumonia or typhoid vaccine, but to select the S. Typhi vector that provides optimal delivery of the PspA antigen in a safe and immunogenic manner.

ELIGIBILITY:
Inclusion criteria:

Subjects will be healthy adults who fully understand the purpose and details of the study.

* Age: 18-40 years inclusive at the time of enrollment
* Sex: Male or non-pregnant female Note: For females, negative pregnancy test at the time of entry. Females agree to use effective birth control measures to prevent pregnancy for one month prior to vaccination and for 28 days after vaccination and while on antibiotics.
* Willing and able to remain in the inpatient facility for the duration of approximately 13-15 days and longer if needed.
* In good health
* Willing and able to provide past medical history
* History of normal,regular bowel habits defined by at least 3 stools per week and less than three stools per day without frequent (greater than one per month) use of laxatives or antidiarrheal agents
* Normal physical examination
* Laboratory evaluation:

Urine dipstick: negative or trace protein Negative urine glucose Complete blood count: WBC, hemoglobin and neutrophil count within normal limits SGPT (ALT) and alkaline phosphatase within normal limits Blood urea nitrogen (BUN), creatinine within normal limits Nonreactive ELISA for HIV-1 Negative HCV-Ab Negative HBSAg Negative nasopharyngeal (a nose and throat swab) culture for S. pneumoniae

* Normal gallbladder ultrasound (ie, no gall stones)
* Able to understand and follow enteric precautions, i.e., practice good hygiene, wash hands thoroughly after using the toilet and avoid food preparation for others until shedding has resolved.
* Lives and works in situations with access to restrooms or bathrooms with flush toilets.
* Willing to avoid eating undercooked poultry and eggs.
* Able to read and willing to sign informed consent form.
* Willing and able to complete a questionnaire to demonstrate an understanding of various protocol issues including potential adverse effects and precautions to limit the spread of Salmonella as discussed in the informed consent.
* Willing and able to undergo rectal swabbing or stool collection.
* Willing and able to maintain a daily memory aid of potential vaccine-associated adverse events, record oral temperatures and collect stool specimens
* Agrees to not be involved in another study during this trial unless discussed with the investigator and approved.

Exclusion criteria:

* History of Salmonella infection or vaccination
* History of pneumococcal vaccine
* Employed as a health care worker with any patient contact, child care provider, long-term care, assisted living or nursing home care taker, or food handler. Has close contact with children less than one year of age, and has close or intimate contact with immunocompromised persons.
* Pregnant or lactating women
* Placement of any prosthetic device of any kind, including but not limited to, orthopedic implants, CNS shunts, endovascular grafts or shunts, cardiac pacemakers, and cochlear implants
* History of splenectomy
* History of gall bladder disease
* History of gastric achlorhydria or use of B12
* Frequent antacid or H2 blocker usage (i.e., Tagamet) (more than once a week)
* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications. [Persons with vitiligo or thyroid disease (e.g. taking thyroid hormone replacement) are not excluded.]
* History of medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol
* History of diarrheal illness within 30 days prior to enrollment (Diarrhea is defined as loose, watery stools occurring more than three times a day lasting more than a day and/or associated with fever.)
* History of anaphylaxis or other serious adverse reactions to vaccines
* History of allergy to ciprofloxacin and quinolones, ampicillin, penicillin, amoxicillin and third generation cephalosporins.
* History of any antibiotic therapy within 14 days prior to vaccination
* Receipt of live attenuated vaccine within 30 days prior to the study
* Receipt of any vaccine within 14 days prior to the study
* Use of experimental agents within 30 days prior to the study
* Receipt of blood products or immune globulin within 6 months prior to the study
* Donation of a unit of blood within 56 days prior to vaccination and for the duration of the study
* Persons taking inhaled steroids will be excluded.
* Persons who required pulsed steroids for conditions other than poison ivy will be excluded.
* Persons who required pulsed steroids for poison ivy within 14 days prior to vaccination will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events, including fever, grade 3 laboratory or systemic AEs, bacteremia, through 6 months), stool cultures and blood cultures | 6 months

SECONDARY OUTCOMES:
Immunogenicity as measured by ELISA (IgA and IgG, PspA , S. Typhi LPS and OMPs) for days 0, 7, 28, 84 and 160 and ELISPOT (IgA PspA , S. Typhi LPS and OMPs) on Days 0 and 7. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Frey, MD, Principal Investigator — Saint Louis University Center for Vaccine Development, St. Louis, MO USA
Locations (1):
- Saint Louis University Center for Vaccine Development, St Louis, Missouri, United States